CLINICAL TRIAL: NCT00814944
Title: A Phase 2, Multi-Center, Randomized, Double-Masked, Placebo-Controlled, Dose-Ranging Clinical Study to Assess the Safety and Efficacy of Subconjunctival Injection of Sirolimus in Patients With Dry Eye in the Controlled Adverse Environmental (CAE) Model
Brief Title: A Dose-Ranging Clinical Study to Assess the Safety and Efficacy of Subconjunctival Injection of Sirolimus in Patients With Dry Eye in the Controlled Adverse Environmental (CAE) Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Collaborators: MacuSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DES-001
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2010-07

CONDITIONS: Dry Eye
Keywords: dry eye; sirolimus; rapamycin
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Group 1 (Experimental)
  Interventions: Drug: Sirolimus
- Dose Group 2 (Experimental)
  Interventions: Drug: Sirolimus
- Dose Group 3 (Experimental)
  Interventions: Drug: Sirolimus
- Dose Group 4 (Placebo Comparator)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Subconjunctival injection of 440 micrograms sirolimus in each eye.
  Other Names: MS-R001, rapamycin
  Arms: Dose Group 2
Drug: Sirolimus — Subconjunctival injection of 220 micrograms sirolimus in each eye.
  Other Names: MS-R003, rapamycin
  Arms: Dose Group 1
Drug: Sirolimus — Subconjunctival injection of 880 micrograms sirolimus in each eye.
  Other Names: MS-R002, rapamycin
  Arms: Dose Group 3
Drug: Sirolimus — Subconjunctival injection of placebo in each eye.
  Arms: Dose Group 4

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an ocular sirolimus (rapamycin) formulation compared to Placebo on the signs and symptoms of dry eye in the CAE Model.

ELIGIBILITY:
Inclusion Criteria include, but are not limited to:

* Have a reported history of dry eye in both eyes;
* Have a history of use of or desire to use an eye drop for dry eye symptoms within the past 6 months.

Exclusion Criteria include, but are not limited to:

* Have contraindications to the use of the study medications;
* Have known allergy or sensitivity to the use of the study medications or diagnostic dyes;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Mean corneal fluorescein staining (inferior region) after CAE exposure. | Day 28
Mean ocular discomfort during CAE exposure. | Day 28

SECONDARY OUTCOMES:
Safety across treatment groups. | Through 28 days
Additional evaluations of dry eye including fluorescein staining, lissamine green staining, conjunctival redness, tear film break-up time, blink rate, ocular protection index, Schirmer's Test, and corneal sensitivity. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Joel Naor, MD, Study Director — MacuSight, Inc.
Locations (1):
- Ophthalmic Research Associates, Andover, Massachusetts, United States